CLINICAL TRIAL: NCT03610022
Title: Study of the Relationship Between the Pharmacokinetics of Vismodegib and Safety Data: a Pilot Study to Therapeutic Optimization in Patients With Basal Cell Carcinoma - OPTIVISMO-1
Brief Title: Relationship Between Pharmacokinetics and Safety of Vismodegib - OPTIVISMO-1
Acronym: OPTIVISMO-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2017/41
Record Dates: First submitted 2018-07-03; First posted 2018-08-01 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Basal Cell Carcinoma; Locally Advanced Basal Cell Carcinoma
Keywords: Vismodegib; Pharmacokinetic; LC-MS/MS-MRM; Human plasma concentrations; Adverse events
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Therapeutics; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with BCC and annexial carcinoma (Experimental): Patients with BCC and annexial carcinoma histologically proven under treatment or new patients under vismodegib
  Interventions: Drug: Treatment with vismodegib

INTERVENTIONS:
Drug: Treatment with vismodegib — Vismodegib 150 mg capsules is administered daily with or without food until disease progression or unacceptable toxicity. Patients are followed in the dermatologic unit of Bordeaux University Hospital (Saint André Hospital) every month. At each consultation, clinical and biological datas, and two blood samples are collected just before taking the drug. One sample is for vismodegib quantification (pharmacokinetic protocol), and the other for the determination of alpha-1 glycoprotein acid level

SUMMARY:
Vismodegib (ERIVEDGE®) at the standard dose of 150 mg/day orally is indicated for the treatment of advanced Basal Cell Carcinoma (BCC) and is associated with many adverse effects. Cramps, alopecia, dysgeusia, weight loss and others observed in clinical practice, compromize compliance and often lead to treatment discontinuation. Currently, it is the only drug available in this indication. Our main objective is to assess the relationship between plasma concentrations of vismodegib, and the occurrence of adverse effects within 6 months of inclusion in the study.

DETAILED DESCRIPTION:
In patients treated with the Hedgehog (Hh) signaling pathway inhibitor, vismodegib, for Basal Cell Carcinoma (BCC), intolerance to this drug is a cause of non-compliance to treatment and often requires therapy discontinuation in spite of its potent anticarcinomic action. Indeed, vismodegib, at the standard dose of 150 mg/day, leads to many heavy side effects often 1 month after therapy initiation. The major side effects are daily or multiple daily cramps (associated with hypometabolism) in 60% of patients, dysgeusia, ageusia and alopecia (related to stem cells), and tiredness. Currently, there is no recommendation for dose adjustment against the occurrence of these adverse effects, so that clinicians propose temporary or definitive therapeutic discontinuation for around 30% of patients. The management of these therapeutic pauses is a challenge for clinicians, as no data are available on their impact on treatment long-term response. We hypothesize that vismodegib side effects are related to high plasma concentrations of drug in many patients. To date, there is no data from phase 3 study, sparse pharmacokinetic data emanating from Phase 1 and 2 studies in various solid tumors.

Patients included are treated with vismodegib (Hedgehog (Hh) pathway inhibitor) for symptomatic metastatic BCC, or for advanced BCC when surgery and radiotherapy are not appropriate. Included patients are new patients initiating a treatment with vismodegib or patients already on vismodegib. The study of the relationship between plasma concentrations of vismodegib and tolerance, requires at each monthly follow-up visits, monitoring of: concentrations of free (unbound to the α1-GPA) and total (bound and unbound) forms of vismodegib, α1-GPA plasma concentrations, patient's status, data on safety and efficacy, and clinical and biological data (covariates that may modulate the vismodegib pharmacokinetics resulting in increased plasma concentrations). Patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BCC and annexial carcinoma histologically proven under treatment or new patients under vismodegib or patients who restarted treatment
* 18 years-old or older
* Complete medical record
* Members or beneficiaries of a social security system,
* Patients must have given informed consent, free and written.

Exclusion Criteria:

* Patients with or without BCC and not treated with vismodegib
* BCC patients who stopped treatment with vismodegib due to non-response or progression on treatment
* Patients under 18 years-old
* Patients whose medical record is incomplete
* Unaffiliated subjects or not beneficiaries of a security system social,
* Patients who have not been informed and have not given their consent, free and written,
* Pregnant and childbearing women without effective contraceptive method
* Patients with confusional state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Serious side effects (grade 2 or more) during the clinical response follow-up to vismodegib | Occurrence from inclusion to 6 months visit
  Patients already on vismodegib will be monitored at inclusion and for 6 months (M0, M1, M2, M3, M4, M5). New patients will be monitored from the end of the first month after inclusion and during 6 months (M1, M2, M3, M4, M5, M6)

SECONDARY OUTCOMES:
Relationship between the plasma concentrations of free and/or total vismodegib, and covariates | From inclusion to 6 months visit
Clinical response to vismodegib in term of efficacy | at least at each visit, from inclusion to 6 months visit
  Classification into 4 categories: progression, stabilité, partial response and complete response according to RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No